CLINICAL TRIAL: NCT01617954
Title: PRospective Study Of MammaPrint in Patients With an Intermediate Recurrence Score
Acronym: PROMIS
Status: Completed | Type: Observational
Sponsor: Agendia (Industry)
Responsible Party: Sponsor
Other Study IDs: PROMIS
Record Dates: First submitted 2012-06-08; First posted 2012-06-13 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Hormone Receptor Positive Malignant Neoplasm of Breast

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients have the option to agree to the storage of excess samples at Agendia.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with MammaPrint Result
  Interventions: Device: MammaPrint

INTERVENTIONS:
Device: MammaPrint — All subjects
  Other Names: 70 gene profile

SUMMARY:
This is a prospective study that will assess the impact of MammaPrint on chemotherapy + endocrine versus endocrine alone treatment decisions in patients with an Oncotype Intermediate Score.

DETAILED DESCRIPTION:
The frequency of chemotherapy + endocrine versus endocrine alone decisions in Oncotype DX intermediate score patients will be calculated before and after receiving the MammaPrint result.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically proven invasive stage I-II, node negative, hormone receptor positive, Her2 negative breast cancer, who received an Oncotype DX intermediate score (18-30)
* ≥ 18 years of age at time of consent
* Written informed consent

Exclusion Criteria:

* Insufficient tissue remaining for Mammaprint FFPE
* Tumor sample shipped to Agendia with ≤ 30% tumor cells or that fails QA or QC criteria
* Women who have started or completed adjuvant chemotherapy or neo-adjuvant chemotherapy

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an Intermediate Recurrence Score
Sampling Method: Probability Sample
Enrollment: 820 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Difference in recommended adjuvant chemotherapy treatment | 30 days
  The frequency of chemotherapy + endocrine versus endocrine alone decisions in Oncotype DX intermediate score patients will be calculated before and after receiving the MammaPrint result. A Chi-square test will be performed for the comparison of the two proportions.

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Tsai, MD, Principal Investigator — Piper Breast Center
Locations (53):
- United States (53):
  - Maricopa Integrated Health System, Phoenix, Arizona
  - Providence Saint Joseph Medical Center, Burbank, California
  - Comprehensive Cancer Center, Palm Springs, California
  - Breastlink, Santa Ana, California
  - Redwood Regional Cancer Center, Santa Rosa, California
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Stamford Hospital, Stamford, Connecticut
  - The Breast Institute at JFK Medical, Atlantis, Florida
  - Halifax Health Center for Oncology, Daytona Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Regional Breast/21st Century Oncology, Fort Myers, Florida
  - Northeast Georgia Cancer Care, Athens, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Loyola University Medical Center, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Delnor Community Hospital, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Orchard Healthcare Research, Northbrook, Illinois
  - CDH Cancer Center, Winfield, Illinois
  - IU Health Bloomington, Bloomington, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Covenant Medical Center, Waterloo, Iowa
  - MedStar Harbor Hospital, Baltimore, Maryland
  - Harry & Jeanette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Western Maryland Health System, Cumberland, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - Mount Auburn Hospital, Cambridge, Massachusetts
  - MetroWest Medical Center, Framingham, Massachusetts
  - St. Vincent Hospital, Worcester, Massachusetts
  - Detroit Clinical Research Center, Detroit, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - St. Louis Cancer Care, Bridgeton, Missouri
  - SSM Cancer Center, St Louis, Missouri
  - Roswell Park Cancer Center, Buffalo, New York
  - North Shore/Monter Cancer Center, Lake Success, New York
  - Columbia University, New York, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - St. Clair Hospital, Pittsburgh, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Knoxville Comprehensive Breast Center, Knoxville, Tennessee
  - Nashville Breast Center, Nashville, Tennessee
  - Texas Health, Dallas, Texas
  - Hematology/Oncology Associates, Alexandria, Virginia
  - Lynchburg Hematology Oncology Clinic, Lynchburg, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Columbia St. Mary's Cancer Center, Milwaukee, Wisconsin
  - Aurora Advanced Healthcare, Milwaukee, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin